CLINICAL TRIAL: NCT03416920
Title: A Smartphone-based Application Post-myocardial Infarction to Manage Cardiovascular Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry); Wellframe, Inc. (Industry)
Responsible Party: Principal Investigator, Pradeep Natarajan, Director of Preventative Cardiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017P002582
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-08

CONDITIONS: Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Enroll and onboard 150 patients with the Wellframe application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellframe (Experimental): Subjects in this arm will use the Wellframe application for 90 days
  Interventions: Other: Wellframe

INTERVENTIONS:
Other: Wellframe — Wellframe mobile phone app

SUMMARY:
The investigators aim to evaluate Wellframe, a patient engagement platform that includes a mobile phone application for patients, for its impact on supporting patients who have undergone a percutaneous coronary intervention. The patient mobile app has articles about cardiovascular disease and other health related topics, patient-reported outcomes surveys, physical activity tracking, reminders for medications and upcoming appointments, and two-way communication with a Wellframe Health Advocate. The Wellframe Health Advocate encourages patients to achieve their health goals and stay engaged in their health. The feasibility of onboarding patients to the app and the clinical efficacy of the platform will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

English-speaking PCI: balloon angioplasty, bare-metal stent, or drug-eluting stent at MGH Smartphone or Tablet (iOS or Android)

Exclusion Criteria:

Recent (within 1mo) illicit substance use or alcohol abuse In-hospital AMI Known pregnancy Dementia or cognitive disability Incarceration

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Natarajan, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetss General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Paruchuri K, Finneran P, Marston NA, Healy EW, Andreo J Jr, Lynch R, Blood AJ, Jones-O'Connor M, Lander B, Kelly N, Vivaldi MT, Traynor K, Wiviott S, Natarajan P. Outcomes of a smartphone-based application with live health-coaching post-percutaneous coronary intervention. EBioMedicine. 2021 Oct;72:103593. doi: 10.1016/j.ebiom.2021.103593. Epub 2021 Oct 14. PMID 34657825

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wellframe
Started | 167
Completed | 118
Not Completed | 49

BASELINE CHARACTERISTICS:
Arm/Group | Wellframe
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 102
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 118

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Readmission at 30 Days
Description: How many subjects were readmitted to the hospital
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Wellframe
Number analyzed (Participants) | 118
Participants | 10

2. Secondary Outcome: Number of Participants With Readmission at 90 Days
Description: How many subjects were readmitted to the hospital
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Wellframe
Number analyzed (Participants) | 118
Participants | 19

3. Secondary Outcome: Number of Participants Enrolled in Clinic-based Cardiac Rehab at 90 Days
Description: Percent of patients discharged after intervention who attend at least one session of clinic-based cardiac rehab
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Wellframe
Number analyzed (Participants) | 118
Participants | 35

ADVERSE EVENTS:
Time Frame: During the study period, 90 days from enrollment.
Description: The number of participants at risk for Other Adverse Events is zero because the study is minimal risk. Since the study involves adding a mobile health component to a treatment plan, risks posed to subjects are similar to those involved with following a post-PCI care plan.
Arm/Group | Wellframe
All-Cause Mortality (participants affected / at risk) | 0/118
Serious Adverse Events (participants affected / at risk) | 0/118
Other Adverse Events (participants affected / at risk) | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT03416920/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT03416920/SAP_001.pdf